CLINICAL TRIAL: NCT06107699
Title: The CHARM Study-Coordinating Transitions from Hospital for Older Adults with Fractures: an Interventional Mixed Methods Study
Brief Title: The CHARM Study-Coordinating Transitions from Hospital for Older Adults with Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horizon Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 101586
Record Dates: First submitted 2023-09-28; First posted 2023-10-30 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Fracture; Frailty; Aging
Keywords: Patient Navigation
MeSH Terms: conditions — Fractures, Bone; Frailty | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Navigator (Experimental)
  Interventions: Other: Patient Navigation
- Standard of Care (No Intervention)

INTERVENTIONS:
Other: Patient Navigation — Assigned a Patient Navigator to provide information on transitional care and community resources.
  Arms: Patient Navigator

SUMMARY:
Background: Fall-related injuries like fractures are on the rise among older adults in New Brunswick. These injuries can lead to hospitalization and adverse health effects. Moreover, transitions from acute care can be complicated and overwhelming, especially for patients and their families. Researching patient navigators as a means of enhancing inpatient care, while also ensuring successful transitions in care for patients, may have positive impacts and help older adults successfully age in place.

Objective: This study seeks to investigate the effects of having support from patient navigators in helping older adults admitted to the Orthopedic Unit with a fracture. Specifically, the objectives are to investigate whether there are differences between patients with patient navigators and those patients receiving standard of care, regarding: the length of stay in acute care; healthcare utilization post-discharge; patient and family experience and satisfaction with care; and, healthcare provider experiences working with patient navigators.

Methods: This study uses a mixed-method concurrent embedded design, in which the quantitative randomized control trial has an embedded qualitative component.

Potential Benefits/Risks: This study is considered low risk. Potential benefits of this study include a better understanding of the impact of support from a patient navigator on inpatient care and patient transitions. This information will be used to inform the development of practical recommendations for policymakers and clinicians on how to enhance inpatient acute care and successful transitions for older adults.

ELIGIBILITY:
Inclusion Criteria: Patients 65 years of age and older admitted to the Orthopedic Unit at SJRH (OU) for a fracture -

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Canadian Patient Experiences Survey Inpatient Care (CPES-IC) | through study completion, 3 months
  Patient satisfaction with care
Healthcare utilization- study specific questionnaire | through study completion, 3 months
Length of stay in acute care | through study completion, 3 months
Global Patient Satisfaction Question- study specific | at study completion, 3 months

SECONDARY OUTCOMES:
Patient experiences- qualitative semi-structured interviews | at study completion, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Hanson, PhD, Study Chair — Horizon Health Network
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanson N, Freeze T, Skerry L, O'Keefe K, Nguyen C, Somal R, Faig K, Jarrett P. Investigating patient navigator impact on older adults' transitions from acute care: A randomized controlled trial with embedded qualitative component. PLoS One. 2026 Feb 4;21(2):e0341251. doi: 10.1371/journal.pone.0341251. eCollection 2026. PMID 41637440